CLINICAL TRIAL: NCT02906072
Title: Effects of an ad Libitum Consumed Low-fat Plant-based Diet Supplemented With Plant-based Meal Replacements on Body Composition Indices
Brief Title: Low Fat Plant-based Diet Effects on Body Composition Indices
Acronym: LFPBDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Jakše s.p. (Other)
Responsible Party: Principal Investigator, Boštjan Jakše, PE teacher, Barbara Jakše s.p.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KR1
Record Dates: First submitted 2016-09-02; First posted 2016-09-19 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Obesity; Weight Loss
Keywords: Obesity; Body fat; Plant-based diet; Plant-based meal replacement
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low fat plant-based diet (Experimental): Low fat plant-based diet with conventional meals and supplemented with plant-based meal replacements and participants attend the lectures on health effects of a low fat plant-based diet.
  Interventions: Behavioral: Low fat plant-based diet; Behavioral: Lectures on health effects of a low fat plant-based diet.
- Control group (Other): Control participants attend the lectures on health effects of a low fat plant-based diet.
  Interventions: Behavioral: Lectures on health effects of a low fat plant-based diet.

INTERVENTIONS:
Behavioral: Low fat plant-based diet — Conventional low fat plant-based meals three times daily. Plant-based meal replacements: Herbalife European Free From vanilla two times daily. Portion sizes and intake is unrestricted.
  Arms: Low fat plant-based diet
Behavioral: Lectures on health effects of a low fat plant-based diet. — Participants attend the lectures on health effects of a low fat plant-based diet.

SUMMARY:
The effect of a diet free from animal-sourced nutrients on body composition in weight reduction programs is not well established. In this non-randomised free living interventional case-control study, the investigators will document the effects of a 10-week, low-fat, plant-based diet supplemented with two daily plant-based meal replacements on body composition indices measured with bioimpedance analysis. Control subjects will be exposed to weekly lectures on the rationale and expected benefits of plant-based nutrition. The investigators hypothesise that low-fat plant based diet supplemented with meal replacements eaten ad libitum allows a significant reduction of body fat without the loss of lean tissue.

DETAILED DESCRIPTION:
This study is designed as a non-randomized, interventional case-control trial, followed by a post-intervention survey of a free living diet optimizing program.

The dietary intervention is executed in free living conditions with participants engaging in their regular daily work and social activities. The plant-based dietary plan includes 3 conventional meals based on starch nutrients (potatoes, sweet potatoes, rice, oatmeal, integral pasta, beans, peas, lentils and similar), fruits (seasonal fruits and various berries) and non-starch vegetables (brassicas, leafy vegetables) and 2 plant based meal replacements. Spices and tomato sauce (without oil) and one regular-sized spoon of flax seed is recommended as well. The participants are recommended to consume no more than 5-6 grams of salt per day. All milk and dairy products, vegetable oils and fats are excluded from the diet. Meat is allowed (but not recommended) once weekly. Two meal replacements are prepared by mixing two scoops of the registered plant-based commercially available nutritional powder (Herbalife European Free From vanilla low GI meal replacement with added plants and herbs, without gluten, lactose or soy, source of protein from pea)) with oat meal and fluid (water or plant milk without oil) thus yielding a 250-400 ml of shake. The total macronutrient composition of the intervention diet is approximated/targeted to 15% protein, 70% carbohydrates and 15% fat. Dietary fibre content is approximated to 40-45 g per day.

No calorie count or limits are instituted to test the hypothesis that ad libitum intake of interventional diet allows significant body fat reduction.

Participants who, after an introductory program presentation, opt not to follow the proposed dietary intervention including meal replacements, but only to attend the lectures on health effects of a low-fat plant-based diet, adjust their diet by their own judgment and attend weekly body composition follow-up measurements, serve as controls.

All participants are followed at weekly intervals. Evaluation of dietary diaries and meal photographs are used to correct and adjust deviations from the targeted dietary plan and to help participants prepare the meals according to the dietary plan. Weekly lectures about the rationale and guidance on attaining the low-fat plant-based diet are given to all subjects (intervention and control group).

Differences between groups will be tested with t-test for unpaired and paired samples, as appropriate. Mann-Whitney and Wilcoxon Signed Rank tests will be used for non-normally distributed data. Chi-square test will be used for categorical variables. Differences between cases and controls will be tested with analysis of covariance (general linear model), with adjustment for baseline variable status, age and sex.

ELIGIBILITY:
Inclusion Criteria:

* Self selected free-living participants older than 18 years of age
* Non overweight, overweight, obese
* Sign informed consent for participation in the study

Exclusion Criteria:

* Pregnant or lactating women, patients with dietary restrictions from a treating physician and patients with active malignant disease are excluded from the study
* Already on plant-based (vegan) diet
* Competitive or top level athletes
* Subjects who take part in any other interventional dietary program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2011-01; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Body fat mass change | Baseline, 10 weeks

SECONDARY OUTCOMES:
Body weight change | Baseline, 10 weeks
Body weight Follow up | Median time lag of 17.4 months
Lean body mass change | Baseline, 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bostjan Jakse, PE teacher, Principal Investigator — Barbara Jakse s.p.

IPD SHARING:
Plan to Share IPD: Yes
Data will be open to public if demanded by the publication/journal.

REFERENCES:
- [Background] Millstein RA. Measuring outcomes in adult weight loss studies that include diet and physical activity: a systematic review. J Nutr Metab. 2014;2014:421423. doi: 10.1155/2014/421423. Epub 2014 Nov 25. PMID 25525513
- [Background] Li Z, Treyzon L, Chen S, Yan E, Thames G, Carpenter CL. Protein-enriched meal replacements do not adversely affect liver, kidney or bone density: an outpatient randomized controlled trial. Nutr J. 2010 Dec 31;9:72. doi: 10.1186/1475-2891-9-72. PMID 21194471
- [Result] Davis LM, Coleman C, Kiel J, Rampolla J, Hutchisen T, Ford L, Andersen WS, Hanlon-Mitola A. Efficacy of a meal replacement diet plan compared to a food-based diet plan after a period of weight loss and weight maintenance: a randomized controlled trial. Nutr J. 2010 Mar 11;9:11. doi: 10.1186/1475-2891-9-11. PMID 20222968
- [Result] Barnard ND, Levin SM, Yokoyama Y. A systematic review and meta-analysis of changes in body weight in clinical trials of vegetarian diets. J Acad Nutr Diet. 2015 Jun;115(6):954-69. doi: 10.1016/j.jand.2014.11.016. Epub 2015 Jan 22. PMID 25620754
- [Derived] Jakse B, Pinter S, Jakse B, Bucar Pajek M, Pajek J. Effects of an Ad Libitum Consumed Low-Fat Plant-Based Diet Supplemented with Plant-Based Meal Replacements on Body Composition Indices. Biomed Res Int. 2017;2017:9626390. doi: 10.1155/2017/9626390. Epub 2017 Mar 28. PMID 28459071